CLINICAL TRIAL: NCT01334554
Title: Effect of Sildenafil Citrate on Insulin Resistance and Endothelial Function in Obese African American Women
Brief Title: Study of Sildenafil Citrate on Insulin Resistance in African American
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Pfizer (Industry)
Responsible Party: Principal Investigator, Cyndya Shibao, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 100713; K23HL103976 (NIH)
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Results first posted 2015-04-10 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: African American; Women; Metabolic Syndrome; Endothelial function; Sildenafil citrate
MeSH Terms: conditions — Metabolic Syndrome; Obesity | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil (Experimental): Sildenafil 20 mg three times a day
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — 20 mg three times a day.
  Other Names: Revatio
  Arms: Sildenafil
Drug: Placebo — No active drug
  Arms: Placebo

SUMMARY:
Obesity has a greater detrimental impact on the health of African American women than on any other racial or gender group. Nearly 80% of African American women are overweight or obese in the United States. Hypertension and insulin resistance are more prevalent among African American women as compared to men and Caucasians. These conditions put them at increased risk for the development of diabetes mellitus and cardiovascular disease.

Recent studies have reported that a substance named Nitric Oxide (NO)may have some beneficial effect on how the body handles blood sugar and blood pressure. Of interest,some studies have shown that African Americans have decreased function of NO in their blood vessels.

In this study proposal the investigators will test if increasing NO function with a PDE-5 inhibitor (sildenafil citrate) will improve pre-diabetes and the health of the inner layer of the blood vessels in obese African American women.

ELIGIBILITY:
Inclusion Criteria:

* Race will be self-defined, but only subjects who report both parents of the same race will be included.
* Age 18-60 years old.
* The investigators will recruit subjects with wide range of BMI 30-45 kg/m2.
* Subjects who have metabolic syndrome or who have a fasting insulin >13. The diagnosis include 3 of the following:

Fasting blood glucose of greater than 100 Triglyceride levels of greater than 150 HDL cholesterol of less than 50 in women Blood pressure of at least 130/85, or on blood pressure medicine Waist girth of more than 35 inches in women. Subjects of childbearing potential will be required to have a negative serum/urine pregnancy test. In addition, they will be asked to use a reliable contraceptive method prior to enrollment as determined by the PI (Dr. Cyndya Shibao).

Exclusion Criteria:

* Previous allergic reactions to any of the study medication (sildenafil) or inability to take study medications as prescribed during the course of the study.
* Type 1 or 2 diabetes mellitus as defined by a fasting glucose of 126 mg/dl or greater.
* Use of antidiabetic medication (insulin, metformin, sulfonylurea, troglitazone)
* Cardiovascular disease such as myocardial infarction within 6 months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (LV hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis or hypertrophic cardiomyopathy.
* Current smokers.
* Significant weight change >5% from baseline in the past three months.
* Pregnancy or breast-feeding.
* History of serious neurological disease such as cerebral hemorrhage stroke, transient ischemic attack.
* History or presence of immunological or hematological disorders.
* Clinical significant gastrointestinal impairment that could interfere with drug absorption.
* Impaired hepatic function (aspartate amino transaminase [AST] and/or alanine amino transaminase [ALT] >1.5X upper limit of normal range).
* Impaired renal function (estimated glomerular filtration rate (eGFR) of <60mL/min).
* Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult.
* History of alcohol or drug abuse.
* Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study.
* Inability to comply with the protocol, e.g. uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study.
* Patients must not be taking nitratest in any form (e.g., nitroglycerin, isosorbide dinitrate, nitroprusside, and others) during this study
* Patients on alpha-blocking drugs (doxazosin, terazosin , or prazosin) will be excluded
* Patients on protease inhibitors (ritonavir and others) will be excluded

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2011-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cyndya Shibao, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marinos A, Celedonio JE, Ramirez CE, Gottlieb J, Gamboa A, Hui N, Yu C, Stein CM, Biaggioni I, Shibao CA. Time-Course Analysis of Flow Mediated Dilation for the Evaluation of Endothelial Function After a High-Fat Meal in African Americans. J Am Heart Assoc. 2015 Nov 5;4(11):e002388. doi: 10.1161/JAHA.115.002388. PMID 26541392

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment started on 03/16/2011 and the first subject was screened on 03/17/2011. Participants were enrolled at Vanderbilt University Medical Center.
Pre-assignment Details: We screened 132 participants. Eighty six participants were excluded because of the following reasons:
  * 80 did not meet inclusion criteria
  * 5 declined to participate after the screening visit
  * 1 excluded because of difficult intravenous access.
Groups:
- Sildenafil: Participants received sildenafil citrate 20 mg three times a day in a fasting condition for 4 weeks
- Placebo: Participants received placebo three times a day for 4 weeks
Period: Overall Study
Arm/Group | Sildenafil | Placebo
Started | 23 | 23
Completed | 19 | 21
Not Completed | 4 | 2
Not completed — Adverse Event | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Sildenafil: Sildenafil 20 mg three times a day for 4 weeks
- Placebo: Placebo three times a day for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Sildenafil | Placebo | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (9.5) | 43 (10.4) | 42.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 164 (5.2) | 162 (4.8) | 163 (5.0)
Weight [Mean (Standard Deviation); unit: kG] | 104.5 (16.7) | 102 (16.4) | 103.3 (16.4)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 39 (5.3) | 39 (5.7) | 39 (5.4)
Waist circumference [Mean (Standard Deviation); unit: cm] | 112 (10.1) | 108 (11.4) | 110 (11.0)
HDL [Mean (Standard Deviation); unit: mg/dL] | 44.0 (9.9) | 45 (11.1) | 44 (10.4)
triglycerides [Mean (Standard Deviation); unit: mg/dL] | 94.0 (52.9) | 85 (48.5) | 89 (50.5)
glucose [Mean (Standard Deviation); unit: mg/dL] | 90 (10.6) | 97 (11.4) | 93.5 (11.4)
insulin [Mean (Standard Deviation); unit: uU/ml] | 15 (7.7) | 14 (9.9) | 14.6 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: insulin sensitivity as measured by frequently sampled intravenous glucose tolerance test
Time Frame: Insulin sensitivity measured at baseline and 4 weeks after the intervention
Measure: Median (Standard Deviation); unit: min-1/pmol/mlx10-5
Groups:
- Sildenafil: Sildenafil: 20 mg TID
- Placebo: Placebo tablets, 1 tablet three times a day
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 19 | 21
min-1/pmol/mlx10-5
  Baseline | 3.4 (2.53) | 2.7 (1.83)
  4-week during intervention | 3.2 (3.02) | 3.0 (2.12)
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; H0= 4-week treatment with sildenafil citrate does not improve insulin sensitivity in obese African American women; Test type: Superiority or Other; p = 0.55, Regression, Linear — p- value was unadjusted. Primary outcome underwent logarithmic transformation; Beta coefficient (linear regression) = 0.12, 95% CI 2-sided [-0.33 to 0.58]

2. Secondary Outcome: Endothelial Function
Description: Endothelial function was measured with flow mediated dilation, percent change
Time Frame: Difference between FMD at baseline and 4 weeks
Population: We detected problems with the ultrasound images obtained to measure flow mediated dilation and therefore only data in 14 subjects in the sildenafil group and in 16 subjects in the placebo were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of brachial artery diameter
Units Other Than Participants: percent change of brachial artery diamet
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 14 | 16
Number analyzed (percent change of brachial artery diamet) | 14 | 16
percentage of brachial artery diameter | 4.7 (2.9) | 5.3 (3.1)
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.649, Regression, Linear — Adjusted for baseline values only; Beta coefficient = 0.46, 95% CI 2-sided [-1.58 to 2.49]

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Sildenafil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 17/23 | 14/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=23) | Placebo (N=23)
Headaches (Nervous system disorders) | 12 (20) | 7 (10)
dizziness (Nervous system disorders) | 5 (6) | 1 (1)
back ache (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
lightheadedness (Nervous system disorders) | 3 (3) | 0 (0)
edema (Musculoskeletal and connective tissue disorders) | 2 (5) | 0 (0)
sinus infection (Ear and labyrinth disorders) | 0 (0) | 2 (2)
flushing (General disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other